CLINICAL TRIAL: NCT01461096
Title: A Randomized, Double-Blinded, Placebo-Controlled, Phase III Trial of the Quadrivalent HPV Vaccine to Prevent Anal Human Papillomavirus Infection in HIV-Infected Men and Women
Brief Title: Quadrivalent HPV Vaccine to Prevent Anal HPV in HIV-infected Men and Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A5298; 11798 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2011-10-26; First posted 2011-10-27 (Estimated); Results first posted 2017-02-07 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quadrivalent HPV Vaccine (Experimental): Participants were prescribed the quadrivalent HPV vaccine at baseline and Weeks 8 and 24.
  Interventions: Biological: Quadrivalent HPV Vaccine
- Placebo Vaccine (Placebo Comparator): Participants were prescribed the placebo vaccine at baseline and Weeks 8 and 24.
  Interventions: Biological: Placebo Vaccine for Male Participants Only; Biological: Placebo Vaccine for Female Participants Only

INTERVENTIONS:
Biological: Quadrivalent HPV Vaccine — Participants were prescribed one intramuscular (IM) injection of the quadrivalent HPV vaccine in the upper arm or thigh at baseline and Weeks 8 and 24.
  Arms: Quadrivalent HPV Vaccine
Biological: Placebo Vaccine for Male Participants Only — Participants were prescribed one IM injection of the placebo vaccine in the upper arm or thigh at baseline and Weeks 8 and 24.
  Arms: Placebo Vaccine
Biological: Placebo Vaccine for Female Participants Only — Participants were prescribed one IM injection of the placebo vaccine in the upper arm or thigh at baseline and Weeks 8 and 24.
  Arms: Placebo Vaccine

SUMMARY:
Men who have sex with men (MSM) have an increased risk of developing anal human papillomavirus (HPV) infections, which can be a risk factor for anal cancer. HIV-infected women are also at risk of anal cancer. This study will evaluate the effectiveness of the Food and Drug Administration (FDA)-approved quadrivalent HPV vaccine, Gardasil, at preventing anal HPV infection in HIV-infected MSM and HIV-infected women.

DETAILED DESCRIPTION:
Anal HPV infection can be a risk factor for anal cancer, which is a common non-AIDS-defining cancer among HIV-infected MSM. Screening for anal cancer is not widely available and can be difficult to implement. People who receive the FDA-approved quadrivalent HPV vaccine, Gardasil, may have a reduced risk of developing anal HPV infection, which may in turn reduce the risk of developing anal cancer. The purpose of this study is to evaluate the effectiveness of the quadrivalent HPV vaccine, Gardasil, at reducing the incidence of anal HPV infections in HIV-infected MSM and HIV-infected women.

This study enrolled HIV-infected MSM and HIV-infected women. Participants were randomly assigned to receive the HPV vaccine or a placebo vaccine. At the screening study visit, participants underwent a physical examination, blood collection, anal swab procedure, oral examination, questionnaires, a high-resolution anoscopy (HRA), and if female, a pregnancy test, vaginal swab, and gynecologic exam. At the entry study visit, participants underwent most of the procedures performed at screening (with the exception of an HRA and a gynecologic exam if female) plus a saliva test. Participants received the HPV vaccine or placebo as an injection into their upper arm or thigh on Day 0 and Weeks 8 and 24. Study staff called participants 2 to 3 days after each vaccination for follow-up monitoring. Additional study visits and procedures occurred at Week 28, Week 52, and every 26 weeks thereafter for at least 3 years and for a maximum of 4 years after the last participant was enrolled in the study. Female participants also had a gynecologic exam at screening, Week 52, and every 52 weeks thereafter; a pregnancy test at screening, baseline, Week 8, Week 24, and as indicated; and self-collected vaginal swabs at screening, entry, Week 28, Week 52, and every 26 weeks thereafter. Peripheral blood mononuclear cells (PBMCs) were collected from some participants at entry, Week 28, and study exit.

The DSMB held a total of four reviews for the study. After careful review of the outcome data in the 4th review held on September 2, 2015, the DSMB commended the study team for a well-run study that provided important results and recommended stopping the study early due to futility. The recommendation was based on meeting the pre-specified criteria for inadequate conditional power to detect a treatment difference at 50% information.

The study was prematurely discontinued on December 31, 2015, which was around eight months earlier than originally planned. With approval from SASC, the study team managed to offer high resolution anoscopy (HRA) procedures to participants whose most recent anal Pap tests showed abnormal results, unless the HRA took place on or after 09/01/14.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load. More information on this criterion can be found in the protocol.
* Laboratory values obtained within 45 days prior to entry by any U.S. laboratory that has a Clinical Laboratory Improvement Amendment (CLIA) certification or its equivalent, or at any network-approved non-U.S. laboratory that operates in accordance with Good Clinical Practices and participates in appropriate external quality assurance programs:

  1. Absolute neutrophil count (ANC) greater than 750 cells/mm^3
  2. Hemoglobin greater than or equal to 9.0 g/dL
  3. Platelet count greater than or equal to 75,000/mm^3
  4. Serum creatinine less than or equal to three times the upper limit of normal (ULN)
  5. Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) less than or equal to five times the ULN
  6. Total or conjugated (direct) bilirubin less than or equal to 2.5 times the ULN
* For men, receptive anal sex (defined as receptive penile-anal sex or receptive oral-anal sex with another man) within 1 year prior to entry
* Anal cytology result from specimen obtained within 45 days prior to entry
* HRA performed within 45 days prior to entry by a certified HRA provider with no evidence of invasive or microinvasive anal cancer by anal biopsy or by visual inspection if no biopsy was obtained. Note: refer to protocol for more information about HRA certification process.
* For women, gynecologic examination (including screening for cervical disease by exfoliative cytology with or without colposcopy) within 45 days prior to entry.
* For women of reproductive potential, a negative serum or urine pregnancy test within 45 days prior to study entry by any U.S. laboratory that has a CLIA certification or its equivalent, or at any network-approved non-U.S. laboratory that operates in accordance with Good Clinical Practices and participates in appropriate external quality assurance programs. More information on this criterion can be found in the protocol.
* Confirmation of the availability of the anal swab, vaginal swab (women only) and Scope oral rinse specimens for HPV DNA PCR obtained at screening. The site must confirm that these samples have been entered into the Laboratory Data Management System (LDMS).
* Ability and willingness of participant or legal representative to provide informed consent

Exclusion Criteria:

* History or current biopsy diagnosis of invasive or microinvasive cancer, i.e.:

  * For all participants: anal or oropharyngeal cancer
  * For men: penile cancer
  * For women: cervical, vulvar, or vaginal cancer
  * More information on this criterion can be found in the protocol.
* Anal, cervical, or vaginal cytological results suspicious for invasive carcinoma at any point prior to entry
* Topical or surgical treatment for intra- or perianal intraepithelial neoplasia or condyloma within 6 months prior to entry. More information on this criterion can be found in the protocol.
* Prior receipt of one or more doses of an HPV vaccine
* Receipt of anticoagulants other than aspirin or nonsteroidal anti-inflammatory drugs (NSAIDS) within 14 days prior to entry
* Known allergy/sensitivity or any hypersensitivity to yeast or any of the components of the study product or its formulation. More information on this criterion can be found in the protocol.
* Active drug or alcohol use or dependence or other condition that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Serious illness requiring systemic treatment and/or hospitalization within 21 days prior to entry
* Hemophilia or other bleeding diatheses
* Use of any systemic antineoplastic or immunomodulatory treatment, systemic corticosteroids other than inhaled corticosteroids or prednisone less than or equal to 10 mg (or equivalent), investigational vaccines, interleukins, interferons, growth factors, or intravenous immunoglobulin (IVIG) within 45 days prior to study entry. NOTE: Routine standard-of-care vaccines (including hepatitis A, hepatitis B, influenza, pneumococcal, and tetanus vaccines) are not exclusionary.
* Expected treatment of hepatitis B or hepatitis C virus with immunomodulatory agents in the 7 months after entry
* Breastfeeding

Min Age: 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 575 (Actual)
Dates: Start 2012-03; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J. Wilkin, MD, MPH, Study Chair — Cornell Clinical Research Site; Ross D. Cranston, MD, Study Chair — University of Pittsburgh Medical Center
Locations (24):
- United States (22):
  - UCLA CARE Center CRS, Los Angeles, California
  - Stanford AIDS Clinical Trials Unit CRS, Palo Alto, California
  - UCSD Antiviral Research Center CRS, San Diego, California
  - Ucsf Hiv/Aids Crs, San Francisco, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Denver Public Health CRS, Denver, Colorado
  - Northwestern University CRS, Chicago, Illinois
  - Rush University CRS, Chicago, Illinois
  - Massachusetts General Hospital CRS (MGH CRS), Boston, Massachusetts
  - Boston Medical Center CRS, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - Weill Cornell Chelsea CRS, New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Columbia P&S CRS, New York, New York
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS, Rochester, New York
  - Chapel Hill CRS, Chapel Hill, North Carolina
  - Cincinnati Clinical Research Site, Cincinnati, Ohio
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - The Miriam Hospital Clinical Research Site (TMH CRS) CRS, Providence, Rhode Island
  - Houston AIDS Research Team CRS, Houston, Texas
- Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Rio de Janeiro, Brazil
- Puerto Rico AIDS Clinical Trials Unit CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] D'Souza G, Wiley DJ, Li X, Chmiel JS, Margolick JB, Cranston RD, Jacobson LP. Incidence and epidemiology of anal cancer in the multicenter AIDS cohort study. J Acquir Immune Defic Syndr. 2008 Aug 1;48(4):491-9. doi: 10.1097/QAI.0b013e31817aebfe. PMID 18614927
- [Background] Piketty C, Selinger-Leneman H, Grabar S, Duvivier C, Bonmarchand M, Abramowitz L, Costagliola D, Mary-Krause M; FHDH-ANRS CO 4. Marked increase in the incidence of invasive anal cancer among HIV-infected patients despite treatment with combination antiretroviral therapy. AIDS. 2008 Jun 19;22(10):1203-11. doi: 10.1097/QAD.0b013e3283023f78. PMID 18525266
- [Background] The DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009).
- [Derived] Kang M, Umbleja T, Ellsworth G, Aberg J, Wilkin T. Effects of Sex, Existing Antibodies, and HIV-1-Related and Other Baseline Factors on Antibody Responses to Quadrivalent HPV Vaccine in Persons With HIV. J Acquir Immune Defic Syndr. 2022 Apr 1;89(4):414-422. doi: 10.1097/QAI.0000000000002891. PMID 34907980
- [Derived] Wilkin TJ, Chen H, Cespedes MS, Leon-Cruz JT, Godfrey C, Chiao EY, Bastow B, Webster-Cyriaque J, Feng Q, Dragavon J, Coombs RW, Presti RM, Saah A, Cranston RD. A Randomized, Placebo-Controlled Trial of the Quadrivalent Human Papillomavirus Vaccine in Human Immunodeficiency Virus-Infected Adults Aged 27 Years or Older: AIDS Clinical Trials Group Protocol A5298. Clin Infect Dis. 2018 Oct 15;67(9):1339-1346. doi: 10.1093/cid/ciy274. PMID 29659751

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In less than 18 months, the full study cohort of 575 participants (472 males and 103 females) were enrolled and randomized in A5298. The first participant was randomized on March 8, 2012 and the last was randomized on August 23, 2013.
Period: Overall Study
Arm/Group | Quadrivalent HPV Vaccine | Placebo Vaccine
Started | 288 | 287
Did Not Start Treatment | 0 | 1 (Randomized but never started treatment and was discontinued from the study)
Completed (Unexpected closure of study. Completed study requirements up to the time of unexpected closure.) | 226 | 226
Not Completed | 62 | 61
Not completed — Death | 3 | 6
Not completed — Severe debilitation, unable to continue | 1 | 1
Not completed — Subj not able to get to clinic | 15 | 13
Not completed — Site is closing | 27 | 30
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Subj not willing to adhere to reqs | 3 | 4
Not completed — Lost to Follow-up | 8 | 4

BASELINE CHARACTERISTICS:
Population: All participants randomized who had results for the respective baseline measure available. The numbers of participants for each measure are shown below.
Groups:
- Total: Total of all reporting groups
Arm/Group | Quadrivalent HPV Vaccine | Placebo Vaccine | Total
Number analyzed (Participants) | 288 | 287 | 575
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 [40 to 52] | 48 [42 to 53] | 47 [41 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 51 | 103
  Male | 236 | 236 | 472
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 125 | 136 | 261
  Black Non-Hispanic | 91 | 89 | 180
  Hispanic (Regardless of Race) | 63 | 54 | 117
  Asian, Pacific Islander | 5 | 7 | 12
  American Indian, Alaskan Native | 2 | 0 | 2
  More than one race | 2 | 1 | 3
Presence of HGAIN at entry [Count of Participants; unit: Participants]
  HGAIN | 95 | 92 | 187
  No HGAIN | 193 | 195 | 388
IV drug history [Count of Participants; unit: Participants]
  Never | 270 | 259 | 529
  Previously | 18 | 28 | 46
HIV RNA results (copies/mL) [Count of Participants; unit: Participants]
  <50 | 226 | 244 | 470
  50-<200 | 23 | 15 | 38
  200-<500 | 13 | 4 | 17
  500-<1000 | 3 | 4 | 7
  1000-<10000 | 10 | 6 | 16
  >=10000 | 7 | 9 | 16
  Missing | 6 | 5 | 11
Lowest documented CD4 count [Median (Inter-Quartile Range); unit: cells/mm^3] — Population: Row population differs from the overall due to Missing
  cells/mm^3
    number analyzed (Participants) | 260 | 255 | 515
    (all) | 254 [105 to 373] | 259 [119 to 419] | 255 [110 to 403]
Absolute CD4 count [Median (Inter-Quartile Range); unit: cells/mm^3] — Population: Row population differs from the overall due to Missing
  cells/mm^3
    number analyzed (Participants) | 285 | 284 | 569
    (all) | 598 [438 to 761] | 614 [435 to 803] | 602 [436 to 767]
Percent CD4 [Median (Inter-Quartile Range); unit: %] — Population: Row population differs from the overall due to Missing
  %
    number analyzed (Participants) | 285 | 284 | 569
    (all) | 32 [25.00 to 38.80] | 31 [23.90 to 37.90] | 31.70 [25 to 38]

OUTCOME MEASURES:

1. Primary Outcome: Time to the First New Persistent Infection of HPV 6, 11, 16, or 18
Description: The outcome for this evaluation was time to the first new persistent infection of any of HPV 6, 11, 16, or 18. Persistent infection was defined as an infection confirmed by positive anal HPV PCR results at 2 consecutive visits at least 16 weeks apart without an intervening negative result. A participant who had a positive measurement on his/her last measurement with no consecutive confirmatory measurement was considered as having a persistent infection. Participants with pre-existing HPV infection at baseline were evaluable for the primary outcome if they were PCR negative for at least one of the four vaccine HPV types at baseline.
  NOTE: Use 5th and 10th percentiles in years from baseline to the first new persistent infection as the summary measure.
Time Frame: From baseline to participant's last study visit, for up to 4 years
Population: The efficacy analysis for persistent anal HPV employed a modified intent-to-treat (mITT) approach wherein all participants who received at least one dose of vaccine and all first new persistent infections that began after the first vaccination were included.
Measure: Number (95.1% Confidence Interval); unit: Years
Arm/Group | Quadrivalent HPV Vaccine | Placebo Vaccine
Number analyzed (Participants) | 286 | 283
Years
  5th percentile | 1.90 [0.94 to 2.46] | 1.04 [0.52 to 2.05]
  10th percentile | 2.92 [2.46 to NA] — Not estimable as the upper limit for survival function at all years was above 90%. | 2.05 [1.94 to 2.95]
Statistical Analysis 1: Comparison: Quadrivalent HPV Vaccine vs Placebo Vaccine; Test type: Superiority or Other; p = 0.350, generalized log-rank test (Sun 1996) — P-value was unadjusted for multiple comparisons and a P-value less than 5% was the threshold for statistical significance; The generalized log-rank test (Sun 1996) was performed to evaluate whether participants in the two arms had the same survival rate; Hazard Ratio (HR) = 0.78, 95.1% CI 2-sided [0.47 to 1.31] — qHPV group represented the numerator for the hazard ratio and Placebo group represented the denominator

2. Secondary Outcome: Number of Participants With Biopsy-proven High-grade Anal Intraepithelial Neoplasia (HGAIN) Occurrences and Reoccurrences After Week 52
Description: HGAIN was defined as AIN2 (moderate dysplasia, with no mention of AIN grade III), AIN3 (severe dysplasia, carcinoma in-situ, or AIN grade II/III), high grade AIN not specified, or adenocarcinoma in situ found in the intra-anal or perianal region.
Time Frame: From Week 52 to participant's last study visit, for up to 4 years
Population: mITT population including all participants who received at least one dose of vaccine.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Vaccine: Participants were prescribed the placebo vaccine at baseline and Weeks 8 and 24.
  Placebo Vaccine for Male Participants Only: Participants were prescribed IM injection of the placebo vaccine in the upper arm or thigh at baseline and Weeks 8 and 24.
  Placebo Vaccine for Female Participants Only: Participants were prescribed one IM injection of the placebo vaccine in the upper arm or thigh at baseline and Weeks 8 and 24.
Arm/Group | Quadrivalent HPV Vaccine | Placebo Vaccine
Number analyzed (Participants) | 288 | 286
Participants | 46 | 45

3. Secondary Outcome: Number of Participants With Anal Cytological Abnormality Occurrences
Description: Anal cytologic abnormalities include: atypical squamous cells undetermined significance (ASCUS), atypical squamous cells favor high-grade SIL/squamous cell carcinoma (ASC-H), low-grade squamous intraepithelial lesion/mild dysplasia/HPV (LSIL), or high-grade SIL/moderate dysplasia to severe dysplasia/carcinoma in situ/features of invasion (HSIL).
Time Frame: At baseline, Week 52, Week 104 and Week 156
Population: mITT population including all participants who received at least one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent HPV Vaccine | Placebo Vaccine
Number analyzed (Participants) | 288 | 286
Participants
  Abnormal cytology at baseline: number analyzed (Participants) | 285 | 284
  Abnormal cytology at baseline | 182 | 188
  Abnormal cytology at Week 52 visit: number analyzed (Participants) | 231 | 229
  Abnormal cytology at Week 52 visit | 123 | 121
  Abnormal cytology at Week 104 visit: number analyzed (Participants) | 199 | 198
  Abnormal cytology at Week 104 visit | 98 | 108
  Abnormal cytology at Week 156 visit: number analyzed (Participants) | 130 | 132
  Abnormal cytology at Week 156 visit | 58 | 72

4. Secondary Outcome: Number of Participants With Grade 3 or 4 Adverse Events (AEs) That Were Possibly, Probably, or Definitely Related to the Vaccine, as Determined by the Local Investigator
Description: To grade diagnoses, signs and symptoms, and laboratory results, sites must refer to the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, august 2009).
Time Frame: From baseline to participant's last study visit, for up to 4 years
Population: mITT population including all participants who received at least one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent HPV Vaccine | Placebo Vaccine
Number analyzed (Participants) | 288 | 286
Participants | 1 | 0

5. Secondary Outcome: Time to First New Persistent Oral HPV Infection of Vaccine Types Detected From Oral Rinse
Description: The outcome for this evaluation was time to the first new persistent infection of any of oral HPV 6, 11, 16, or 18. Persistent infection was defined as an infection confirmed by positive oral HPV PCR results at 2 consecutive visits at least 16 weeks apart without an intervening negative result. A participant who had a positive measurement on his/her last measurement with no consecutive confirmatory measurement was considered as having a persistent infection. Participants with pre-existing HPV infection at baseline were evaluable for the primary endpoint if they were PCR negative for at least one of the four vaccine HPV types at baseline.
  NOTE: Use 5th and 10th percentiles in years from baseline to the first new persistent infection as the summary measure.
Time Frame: From baseline to participant's last study visit, for up to 4 years
Population: mITT population wherein all participants who received at least one dose of vaccine and all first new persistent infections that began after the first vaccination were included.
Measure: Number (95.1% Confidence Interval); unit: Years
Arm/Group | Quadrivalent HPV Vaccine | Placebo Vaccine
Number analyzed (Participants) | 288 | 286
Years
  5th percentile | NA [2.99 to NA] — Not estimable as the estimate for survival function at all years was above 95%. (Note: A total of 7 events were observed, and the 3-year persistent infection free rate was about 0.97.) | NA [1.90 to NA] — Not estimable as the estimate for survival function at all years was above 95%. (Note: A total of 10 events were observed, and the 3-year persistent infection free rate was about 0.96.)
  10th percentile | NA [NA to NA] — Not estimable as the estimate for survival function at all years was above 90%. | NA [NA to NA] — Not estimable as the estimate for survival function at all years was above 90%.

ADVERSE EVENTS:
Time Frame: From baseline to participant's last study visit, for up to 4 years
Description: At entry, the protocol required reporting of signs/symptoms >=Grade 3 that occurred within 14 days before entry. After entry, the protocol required reporting of signs/symptoms >=Grade 3, laboratory results >=Grade 3 and events that led to a change in treatment, regardless of grade. HGB, PLT, ANC, AST, ALT, INR, total and direct bilirubin, creatinine were reported regardless of grade. The DAIDS AE Grading Table (V1.0) and Expedited AE Manual (V2.0) were used.
Groups:
- qHPV: Participants were prescribed the quadrivalent HPV vaccine at baseline and Weeks 8 and 24.
  Quadrivalent HPV Vaccine: Participants were prescribed one intramuscular (IM) injection of the quadrivalent HPV vaccine in the upper arm or thigh at baseline and Weeks 8 and 24.
- Placebo: Participants were prescribed the placebo vaccine at baseline and Weeks 8 and 24.
  Placebo Vaccine for Male Participants Only: Participants were prescribed one IM injection of the placebo vaccine in the upper arm or thigh at baseline and Weeks 8 and 24.
  Placebo Vaccine for Female Participants Only: Participants were prescribed one IM injection of the placebo vaccine in the upper arm or thigh at baseline and Weeks 8 and 24.
Arm/Group | qHPV | Placebo
All-Cause Mortality (participants affected / at risk) | 3/288 | 6/287
Serious Adverse Events (participants affected / at risk) | 33/288 | 46/287
Other Adverse Events (participants affected / at risk) | 87/288 | 95/287
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | qHPV (N=288) | Placebo (N=287)
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Abdominal mass (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 2
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 3
Chest pain (General disorders) | 2 | 5
Death (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 1 | 0
Chlamydial infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 2 | 2
Meningitis viral (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 1
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 3
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Primary syphilis (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Scrotal abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 3
Viral infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Stab wound (Injury, poisoning and procedural complications) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Follicle centre lymphoma diffuse small cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 2
Acute psychosis (Psychiatric disorders) | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Substance abuse (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 1
Genital ulceration (Reproductive system and breast disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Intervertebral disc operation (Surgical and medical procedures) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | qHPV (N=288) | Placebo (N=287)
Abdominal pain (Gastrointestinal disorders) | 13 | 16
Anogenital dysplasia (Gastrointestinal disorders) | 11 | 20
Diarrhoea (Gastrointestinal disorders) | 16 | 26
Nausea (Gastrointestinal disorders) | 16 | 20
Vomiting (Gastrointestinal disorders) | 7 | 20
Chills (General disorders) | 21 | 17
Fatigue (General disorders) | 18 | 19
Pyrexia (General disorders) | 31 | 30
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 | 19
Headache (Nervous system disorders) | 16 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 33 | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 20
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 18 | 14
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 19 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights